CLINICAL TRIAL: NCT06032234
Title: Development and Evaluation of a Web-based Diet Quality Screener for Vegans (VEGANScreener)
Acronym: VEGANScreener
Status: Completed | Type: Observational
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Berner Fachhochschule (Unknown)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Principle Investigator, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: VEGANScreenerCH
Record Dates: First submitted 2023-08-25; First posted 2023-09-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and saliva samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Omnivorous: Participants following an omniviours diet
  Interventions: Other: This is an observational study
- Vegan: Participants following a vegan diet
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study — This is an observational study

SUMMARY:
The primary objective of this study is to assess the construct validity and criterion validity for associations of the VEGANScreener with nutrient intakes from reference methods and associations with biomarkers of dietary intake. The investigators hypothesize that the screener is a valid tool to assess diet quality in the vegan population. The study will assess construct validity by testing whether the measure relates as it should to other measures (e.g., age, gender, education, SES differences).

The investigators will assess concurrent and predictive validity (types of criterion validity) by evaluating associations and agreement between 'gold standards', such as diet records, biomarkers, and multi-metabolite signatures of intake. The investigators will examine associations of vegan diet quality with biomarkers of nutritional status, biomarkers of disease, and anthropometric measures and hypothesize that a higher diet quality in vegans is associated with a more favourable profile among vegans, for example, a lower blood pressure. This study is part of the European VEGANScreener Consortium.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported vegans (≥2 years on a vegan diet; vegan diet defined as not consuming any dietary animal products more often than once/month, honey excluded)
2. Self-reported omnivores. Consuming on average daily (at least 5 times/week) meat/meat products.
3. Age 18 to 65 years (1:1 ratio 18-35,99 and 36-65)
4. Males and females (1:1 ratio)

Exclusion Criteria:

1. Self-identified pescatarians (excluding all meat, except for fish/seafood) and reductarians/flexitarians (intentionally reducing intake of animal-based products)
2. History of a disease known to affect intermediary metabolism (e.g., any diabetes on treatment, i.e. medication or lifestyle recommendations, thyreopathies, cancer etc.)
3. BMI>30 kg/m2
4. History of disease of intestinal integrity (i.e., inflammatory bowel disease, chronic pancreatitis, other malabsorption, etc.).
5. Pregnant or breastfeeding females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — An equal number of male and female participants will be included. Inclusion is based on self-representation of gender identity.
Study Population: Healthy participants following a vegan or omnivours diet (ratio 1:1).
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Validity of the vegan screener | Baseline
  The validity will be assessed by calculating associations between the screener and reference method.

SECONDARY OUTCOMES:
Dietary intake | Baseline
  Dietary intake will be assessed using a weighed food record
Food habits | Baseline
  Food habits will be assessed using a food frequency questionnaire
Vitamin D status | Baseline
  Vitamin D status will be measured from venous blood samples
Homocysteine status | Baseline
  Homocysteine will be measured from venous blood samples
holo-transcobalamin | Baseline
  holo-transcobalamin will be measured from venous blood samples
Methoylmalonic acid | Baseline
  Methoylmalonic acid will be measured from venous blood samples
Vitamin B2 status | Baseline
  Vitamin B2 will be measured from venous blood samples
Vitamin C status | Baseline
  Vitamin C will be measured from venous blood samples
Folic acid status | Baseline
  Folic acid will be measured from venous blood samples
Magnesium status | Baseline
  Magnesium status will be determined from venous blood samples
Zinc status | Baseline
  Zinc status will be determined from venous blood samples
Selenoprotein-P status | Baseline
  Selenoprotein-P status will be determined from venous blood samples
Ferritin concentration | Baseline
  Ferritin concentration will be determined from venous blood samples
Soluble transferrin receptor concentration | Baseline
  Soluble transferrin receptor will be determined from venous blood samples
Hemoglobin concentration | Baseline
  Hemoglobin will be determined from venous blood samples
Creatinine concentration | Baseline
  Creatinine will be determined from venous blood samples
Uric acid concentration | Baseline
  Uric acid will be determined from venous blood samples
Urea concentration | Baseline
  Urea will be determined from urine samples samples
Iodine concentration | Baseline
  Iodine status will be determined from urine samples samples
Potassium concentration | Baseline
  Potassium status will be determined from urine samples samples iodine, potassium, sodium, calcium, creatinine)
Sodium concentration | Baseline
  Sodium status will be determined from urine samples samples
Calcium concentration | Baseline
  Calcium status will be determined from urine samples samples i
Creatinine concentration | Baseline
  Creatinine will be determined from urine samples samples
C-reactive protein concentration | Baseline
  The inflammatory marker hsCRP will be determined from serum
Triglyceride concentration | Baseline
  Triglyceride concentration will be determine from venous blood samples
Free fatty acid concentration | Baseline
  Free fatty acid concentration will be determine from venous blood samples (
Eicosapentanoic acid | Baseline
  Eicosapentanoic acid (in % of total FA) will be determine from venous blood samples
Docosahexanoic acid | Baseline
  Docosahexanoic acid (in % of total FA) will be determine from venous blood samples
LDL-cholesterol concentration | Baseline
  LDL-cholesterol concentration will be determine from venous blood samples
HDL-Cholesterol concentration | Baseline
  HDL-Cholesterol concentration will be determine from venous blood samples
Cholesterol concentration | Baseline
  Cholesterol concentration will be determine from venous blood samples
Glucose concentration | Baseline
  Glucose will be measured from venous blood samples
Well being questionnaire | Baseline
  Participants well being will be assessed using a questionnaire. The scale of each question ranges from 0 to 10, 10 representing the highest well being
VEGANScreener | Baseline and day 2
  The VEGANScreener assesses diet quality using 29 questions of frequency of consumption of different foods and food groups.
Weight | Baseline
  Weight will be measured in kg
Height | Baseline
  Height will be measured in m
Waist circumference | Baseline
  Waist circumference will be measured in cm
Hip circumference | Baseline
  Hip circumference will be measured in cm

OTHER OUTCOMES:
International Physical Activity Questionnaire iPAQ | Baseline
  Physical activity will be assessed using a questionnaire using the iPAQ
Blood pressure | Baseline
  Systolic and diastolic blood pressure will be measured
Heart rate | Baseline
  Heart rate will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Canton of Zurich, Switzerland